CLINICAL TRIAL: NCT05858723
Title: Allergic Contact Dermatitis to Hydroperoxides of Linalool - a Repeated Open Application Test (ROAT) Study
Brief Title: Repeated Open Application Test (ROAT) Study With Hydroperoxides of Linalool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Allergy Research Center, Denmark (Other)
Responsible Party: Principal Investigator, Sofia Hedvig Christina Botvid, M.D, Ph.D. fellow, National Allergy Research Center, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-23018400
Record Dates: First submitted 2023-05-02; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Patch Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allergic participants (Experimental)
  Interventions: Diagnostic Test: ROAT
- Healthy participants (Experimental)
  Interventions: Diagnostic Test: ROAT

INTERVENTIONS:
Diagnostic Test: ROAT — Repeated Open Application Test
  Other Names: Patch testing and punch biopsies

SUMMARY:
Linalool is currently one of the most used fragrance substances in cosmetic and household products. Previous studies report a high prevalence (5.9-11.7%) of contact allergy to hydroperoxides of linalool (Lin-OOH)1.0% in pet. among patch tested patients. The optimal test concentration of Lin-OOH in patch tests is not known and requires further investigation. It is of great importance to establish the optimal test concentration and elicitation threshold of Lin-OOH to improve diagnosis and prevent development of Allergic Contact Dermatitis (ACD).

We want to mimic real-life exposure to Lin-OOH, by conducting a ROAT (Repeated Open Application Test) study, on 40 adult participants (20 patients with confirmed contact allergy to Lin-OOH, and 20 healthy participants) to low doses of Lin-OOH using a simulated "perfume", during a maximum of 21 days of exposure.

With this knowledge, we aim to:

1. Establish the optimal patch test concentration to diagnose ACD to Lin-OOH
2. In case of confirmed contact allergy, examine the threshold value for the development of ACD upon daily exposure to a simulated leave-on cosmetic product

ELIGIBILITY:
Allergic participants:

1. Inclusion criteria

   * Positive (at least one reading) or doubtful patch test (at least two readings) result to hydroperoxides of Linalool within the last ten years
   * Aged 18 years or older
   * Received written and verbal information of the study
   * Signed written consent form
2. Exclusion criteria

   * Active eczema in test areas (volar forearms)
   * Pregnancy or breast feeding
   * Treatment with topical corticosteroids or other immune suppressants on/near test areas within two weeks prior to study start
   * Systemic immune-suppressant treatment within seven days prior to study start
   * UV exposure of test areas within three weeks prior to study start
   * Unable to cooperate or communicate with the investigators

Healthy controls:

1. Inclusion criteria

   * Aged 18 years or older
   * Received written and verbal information of the study
   * Signed written consent form
2. Exclusion criteria

   * Known or possible contact allergy to hydroperoxides of Linalool
   * Known contact allergy to other fragrance allergens
   * Active eczema or other known relevant skin diseases
   * Pregnancy or breast feeding
   * Treatment with topical corticosteroids or other immune suppressants on/near test areas within four weeks prior to study start.
   * Systemic immune-suppressant treatment within four weeks prior to study start.
   * UV exposure of test areas within three weeks prior to study start.
   * Participation in other clinical studies within four weeks prior to study start.
   * Unable to cooperate or communicate with the investigators.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Establish the optimal patch test concentration to diagnose allergic contact dermatitis to hydroperoxides of linalool via a Repeated Open Application Test | 6 months
  Establish the optimal patch test concentration to diagnose allergic contact dermatitis to hydroperoxides of linalool via Repeated Open Application Test
In case of confirmed contact allergy, examine the threshold value for the development of ACD upon daily exposure to a simulated leave-on cosmetic product | 6 months
  In case of confirmed contact allergy, examine the threshold value for the development of ACD upon daily exposure to a simulated leave-on cosmetic product

SECONDARY OUTCOMES:
The Lin-OOH chemicals can penetrate the skin barrier and reside in the local skin tissue | 12 months
  Chemical analysis of skin punch biopsies from the exposed skin of the patients' lower back: time of flight secondary ion mass spectrometry (ToF-SIMS) analysis of Lin-OOH in the skin.

IPD SHARING:
Plan to Share IPD: No